CLINICAL TRIAL: NCT03386487
Title: A Phase 2B, 8-week, Randomized, Double-Blind, Placebo-Controlled, Parallel Study to Evaluate Efficacy, Safety and Tolerability of the Fatty Acid Amide Hydrolase (FAAH) Inhibitor PF-04457845 in Adults With DSM5 Current Cannabis Use Disorder (CUD)
Brief Title: Fatty Acid Amide Hydrolase (FAAH) Inhibitor Treatment of Cannabis Use Disorder (CUD)
Acronym: FAAH-I MULTI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Columbia University (Other); Johns Hopkins University (Other); Medical University of South Carolina (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000022450; 1U01DA045372-01 (NIH)
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Cannabis Use Disorder
MeSH Terms: interventions — N-pyridazin-3-yl-4-(3-((5-(trifluoromethyl)pyridin-2-yl)oxy)benzylidene)piperidine-1-carboxamide

STUDY DESIGN:
Intervention Model Description: Phase 2B
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-04457845 (Active Comparator): Subjects will be randomized to Fatty Acid Amide Hydrolase (FAAH) Inhibitor; 4 mg PF-04457845 QD x 8 weeks
  Interventions: Drug: PF 04457845
- Placebo (Placebo Comparator): Subjects will be randomized to placebo
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: PF 04457845 — Study medication will be administered at 4mg by mouth daily for eight weeks.
  Arms: PF-04457845
Drug: Placebo Oral Tablet — Placebo comparator will be administered by mouth daily for eight weeks.
  Arms: Placebo

SUMMARY:
A Phase 2B, 8-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy, Safety and Tolerability of the Fatty Acid Amide Hydrolase (FAAH) Inhibitor PF-04457845 in Adults with DSM-5 Current Cannabis Use Disorder (CUD)

DETAILED DESCRIPTION:
The efficacy, safety and tolerability of the FAAH Inhibitor PF-0447845 in reducing cannabis use will be studied in a 4-site randomized, double-blind, placebo-controlled, parallel-group, outpatient clinical trial comparing PF-04457845 (4mg) and placebo in DSM-5 CUD individuals. Participants will be randomized in a 1:1 ratio to either PF-04457845 or placebo using random block sizes of 2 and 4, stratified by site and degree of cannabis use. Participants will receive motivational interviewing for 2 weeks before being randomized to receive study medication to make a quit attempt within the first week of treatment. Participants will receive active or placebo PF-04457845 for 8 weeks during which time they will be evaluated weekly in face to face visits. In addition, daily assessment of adherence to study medication and cannabinoid use will be conducted daily by cellphone. Measures of cannabinoid exposure (self-reported and urine toxicology), and problems related to the use of cannabis, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-60 years, inclusive.
2. Male or Female.
3. Individuals with DSM-V criteria for Cannabis Use Disorder .
4. Positive for urinary THC-COOH at both screening visits.
5. Must express a willingness at screening to set a date within the first week of randomization to attempt to quit using cannabis.

Exclusion Criteria:

1. Clinically significant unstable medical disorders (as determined by the site investigator).
2. Laboratory tests with clinically significant abnormalities (as determined by the site investigator)
3. Pregnancy by history and or laboratory confirmation (serum HCG).
4. Lactation.
5. Physiological dependence on another substance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 228 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak C D'Souza, MD, Principal Investigator — Yale University
Locations (4):
- United States (4):
  - Connecticut Mental Health Center, New Haven, Connecticut
  - Johns Hopkins University, Baltimore, Maryland
  - Columbia University Medical College / New York State Psychiatric Institute, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PF-04457845 | Placebo
Started | 116 | 112
Completed | 89 | 91
Not Completed | 27 | 21
Not completed — Lost to Follow-up | 5 | 6
Not completed — Withdrawal by Subject | 11 | 7
Not completed — Physician Decision | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04457845 | Placebo | Total
Number analyzed (Participants) | 116 | 112 | 228
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 116 | 112 | 228
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.48 (10.32) | 32.91 (10.52) | 32.18 (10.42)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 68 | 75 | 143
  Female | 47 | 37 | 84
  Transgender | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 16 | 36
  Not Hispanic or Latino | 96 | 96 | 192
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 47 | 53 | 100
  White | 47 | 45 | 92
  More than one race | 13 | 9 | 22
  Unknown or Not Reported | 6 | 1 | 7
Marital Status [Count of Participants; unit: Participants]
  Married | 16 | 20 | 36
  In a Relationship & Living Together | 12 | 10 | 22
  In a Relationship | 10 | 10 | 20
  Divorced or Annulled | 7 | 5 | 12
  Separated | 4 | 4 | 8
  Single | 45 | 40 | 85
  Never Married | 22 | 23 | 45
Education [Count of Participants; unit: Participants]
  Less than High School Diploma | 4 | 3 | 7
  High School Diploma | 24 | 24 | 48
  GED | 6 | 6 | 12
  Some College | 29 | 33 | 62
  Associates Degree | 15 | 10 | 25
  Bachelors Degree | 28 | 27 | 55
  Masters Degree | 7 | 8 | 15
  Professional / Doctoral Degree | 3 | 1 | 4
Employment Status [Count of Participants; unit: Participants]
  Full-Time Job | 54 | 44 | 98
  Part-Time Job | 29 | 30 | 59
  Temporarily Laid Off, On Leave | 3 | 1 | 4
  Looking for Work, Unemployed | 13 | 18 | 31
  Retired | 1 | 2 | 3
  Disabled, Permanently/Temp | 0 | 1 | 1
  Keeping House | 0 | 2 | 2
  Student | 7 | 5 | 12
  Other | 9 | 9 | 18
Cannabis Use Severity (CUD) [Count of Participants; unit: Participants] — Cannabis use disorder (CUD) is a diagnosis from the DSM V is based on 11 criteria or symptoms. The severity of the person's problems can be categorized as: Mild (two to three symptoms), Moderate (four to five symptoms), Severe (six or more symptoms).
  Participants
    Moderate | 63 | 60 | 123
    Severe | 53 | 52 | 105

OUTCOME MEASURES:

1. Primary Outcome: Time Line Follow Back (TLFB) for Cannabis Use
Description: Change in the average number of times per day of self-reported cannabis consumption measured by the Timeline Follow Back approach for Cannabis Use in which participants quantify and report their frequency of cannabis use prior to study participation and throughout the study. Differences between groups in the change from baseline use (2 weeks prior to randomization) in the average number of times per day of self-reported consumption of cannabis or a cannabis containing product in the last 4 weeks of treatment captured using the daily TLFB data collected during CAROMA calls.
Time Frame: Change from baseline in self reported cannabis use as measured by the TLFB approach at baseline and then weekly average daily use over 8 weeks.
Measure: Mean (Standard Deviation); unit: times/day of self-reported cannabis use
Arm/Group | PF-04457845 | Placebo
Number analyzed (Participants) | 105 | 109
times/day of self-reported cannabis use
  Week 1 | 1.921 (1.538) | 1.768 (1.758)
  Week 2 | 1.201 (1.638) | 1.066 (1.702)
  Week 3 | 1.308 (1.881) | 1.06 (1.663)
  Week 4 | 1.316 (1.956) | 0.998 (1.414)
  Week 5 | 1.234 (1.8) | 1.214 (2.22)
  Week 6 | 1.252 (1.639) | 1.079 (1.645)
  Week 7 | 1.321 (1.762) | 0.91 (1.3)
  Week 8 | 1.113 (1.481) | 0.936 (1.417)

2. Primary Outcome: Urinary Levels of THC-COOH (ng/ml)
Description: Assay of the levels of the principal metabolite of THC (THC-COOH) in urine samples at baseline and bi-weekly over 8 weeks.
Time Frame: baseline, week 1, week 3, week 5, week 7, and week 9 visits
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | PF-04457845 | Placebo
Number analyzed (Participants) | 106 | 106
ng/ml
  Screening | 5.959 (6.633) | 5.571 (6.542)
  Week 1 | 5.077 (4.837) | 5.747 (7.456)
  Week 3 | 3.069 (3.385) | 3.92 (6.673)
  Week 5 | 3.482 (5.064) | 4.465 (7.411)
  Week 7 | 3.241 (5.67) | 4.223 (7.724)
  Week 9 | 3.222 (3.913) | 3.952 (7.511)

ADVERSE EVENTS:
Time Frame: The adverse events reported were collected throughout the treatment phase of the study (randomization to the end of week 8; i.e. the beginning of the treatment phase of the study through the end of the treatment phase of the study).
Arm/Group | PF-04457845 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/112
Serious Adverse Events (participants affected / at risk) | 2/116 | 0/112
Other Adverse Events (participants affected / at risk) | 89/116 | 91/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04457845 (N=116) | Placebo (N=112)
Abscess Removal (General disorders) | 1 | 0
Bowel Obstruction (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04457845 (N=116) | Placebo (N=112)
Tachycardia (Cardiac disorders) | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 1 | 2
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1
Hordeolum (Eye disorders) | 0 | 1
Lacrimation Increased (Eye disorders) | 0 | 1
Vision Blurred (Eye disorders) | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 4 | 2
Abdominal Distension (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 4 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 8 | 7
Bruxism (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 8
Dry Mouth (Gastrointestinal disorders) | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 6
Flatulence (Gastrointestinal disorders) | 1 | 1
Frequent Bowel Movements (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 15 | 16
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Salivary Hypersecretion (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 8 | 8
Asthenia (General disorders) | 1 | 2
Blue Tongue (General disorders) | 1 | 0
Chills (General disorders) | 4 | 0
Chest Discomfort (General disorders) | 4 | 1
Chest Pain (General disorders) | 0 | 2
Energy Increased (General disorders) | 0 | 2
Fatigue (General disorders) | 6 | 7
Feeling Abnormal (General disorders) | 1 | 2
Flushing (General disorders) | 1 | 0
Hyperhidrosis (General disorders) | 6 | 3
Hot Flush (General disorders) | 0 | 3
Lethargy (General disorders) | 1 | 0
Night Sweats (General disorders) | 3 | 3
Peripheral Swelling (General disorders) | 1 | 0
Puncture site bruise (General disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 4
Thirst (General disorders) | 1 | 0
Hypoergia (Immune system disorders) | 0 | 1
Rhinitis allergic (Immune system disorders) | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 2 | 3
Sinusitis (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Herpes Simplex (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 2
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Toenail Laceration (Injury, poisoning and procedural complications) | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1
Retinal Detachment (Injury, poisoning and procedural complications) | 1 | 0
Lump on Right Side of Chest (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin Increased (Investigations) | 2 | 0
Blood Glucose Increased (Investigations) | 0 | 1
Blood Pressure Increased (Investigations) | 0 | 1
Elevated Absolute Eosinophils (Investigations) | 0 | 1
Heart Rate Increased (Investigations) | 0 | 1
Hepatic Enzyme Increased (Investigations) | 1 | 0
Transaminitis (Investigations) | 1 | 0
Weight Decreased (Investigations) | 0 | 2
Weight Increased (Investigations) | 1 | 1
Hyperphagia (Metabolism and nutrition disorders) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 14 | 12
Increased Appetite (Metabolism and nutrition disorders) | 6 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Food Craving (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Hand Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Ligament Sprain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle Strain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Abnormal Dreams (Nervous system disorders) | 17 | 19
Ageusia (Nervous system disorders) | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1
Balance Disorder (Nervous system disorders) | 0 | 1
Disorientation (Nervous system disorders) | 0 | 1
Disturbance in Attention (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 15 | 5
Headache (Nervous system disorders) | 24 | 26
Hypersomnia (Nervous system disorders) | 0 | 2
Improved Sleep (Nervous system disorders) | 0 | 1
Initial Insomnia (Nervous system disorders) | 8 | 2
Insomnia (Nervous system disorders) | 17 | 19
Lethargy (Nervous system disorders) | 0 | 1
Memory Impairment (Nervous system disorders) | 0 | 2
Migraine (Nervous system disorders) | 0 | 1
Poor Quality Sleep (Nervous system disorders) | 4 | 9
Paraesthesia (Nervous system disorders) | 0 | 1
Restlessness (Nervous system disorders) | 2 | 2
Sedation (Nervous system disorders) | 1 | 0
Sleep Paralysis (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 4 | 11
Tremor (Nervous system disorders) | 0 | 3
Agitation (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 16 | 14
Apathy (Psychiatric disorders) | 1 | 1
Clearheaded (Psychiatric disorders) | 1 | 0
Dissociative State (Psychiatric disorders) | 0 | 1
Disturbed Thinking in Context of Cannabis Intoxication (Psychiatric disorders) | 0 | 1
Depressed Mood (Psychiatric disorders) | 16 | 6
Depressive Symptoms (Psychiatric disorders) | 1 | 1
Euphoric Mood (Psychiatric disorders) | 2 | 2
Flashes (Psychiatric disorders) | 0 | 1
Hypomania (Psychiatric disorders) | 0 | 1
Internal feeling of being high without using THC (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 19 | 17
Mood Swings (Psychiatric disorders) | 1 | 1
Nightmare (Psychiatric disorders) | 0 | 2
Panic Attack (Psychiatric disorders) | 2 | 2
Paranoia (Psychiatric disorders) | 1 | 0
Slight Increase in Alcohol Use (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 2 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 1
Cystitis (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1
Pyelonephritis (Renal and urinary disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 2
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 1 | 0
Intermenstrual Bleeding (Reproductive system and breast disorders) | 2 | 0
Libido Decreased (Reproductive system and breast disorders) | 1 | 1
Nocturnal Emission (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal Swelling (Reproductive system and breast disorders) | 1 | 0
Aphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
COVID-19 Positive (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Paraesthesia (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 4
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Sunburn (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT03386487/Prot_SAP_000.pdf